CLINICAL TRIAL: NCT02462005
Title: Ranger DEB All Comers Registry - Treatment of Femoro-popliteal Atherosclerotic Lesions Using the Ranger Paclitaxel Coated Balloon Catheter: An All Comers Registry.
Brief Title: Treatment of Femoro-popliteal Atherosclerotic Lesions Using the Ranger Paclitaxel Coated Balloon Catheter. All Comers Registry.
Status: Completed | Type: Observational
Sponsor: Klinikum Arnsberg (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Ranger SFA Registry
Record Dates: First submitted 2015-05-27; First posted 2015-06-03 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Atherosclerotic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ALL COMERS: Patients implanted or scheduled for an implant with a Ranger Drug coated balloon.

SUMMARY:
A total of up to 250 patients from an all-comers patient population with infrainguinal atherosclerotic disease who are implanted or scheduled for an implant with a Ranger Drug coated balloon.

Interim analysis will be carried out for every 50 subjects enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Patient must be willing to sign a a patient informed consent form.
* Patient with de novo, restenotic or reoccluded lesions in the infrainguinal .arteries implanted or scheduled for an implant with a Ranger Drug coated balloon.
* Target vessel reference diameter 2.5 to 8 mm.

Exclusion Criteria:

* Subjects pregnant or planning to become pregnant during the course of the study.
* Life expectancy of less than 1 year.
* Known allergy to concomitant medication, contrast agents (that cannot be medically managed), anti-platelet, anti-coagulant or thrombolytic medications. Subject enrolled in another study that has not reached its primary endpoint at the time of enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from an all-comers patient population with infrainguinal atherosclerotic disease who are implanted or scheduled for an implant with a Ranger Drug coated balloon and who fulfill the in/exclusion criteria at approved investigational centres are eligible for participation in the Ranger DEB-Comers Registry.
Sampling Method: Non-Probability Sample
Enrollment: 171 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Clinical primary endpoint: Major Adverse Events (MAE) defined as composite of freedom from device- and procedure-related mortality through 30 days, freedom from major target limb amputation and TLR within 6 months post-index procedure. | 6 Months
Performance primary endpoint: Primary patency at 12 months, defined as freedom from > 50% restenosis with no clinically-driven reintervention | 12 Months

SECONDARY OUTCOMES:
Primary patency at 6 and 24 months, defined as freedom from > 50% restenosis with no clinically-driven reintervention | 6 and 24 Months
MAE at 12 and 24 months | 12 and 24 Months
Technical success, defined as successful vascular access and completion of the endovascular procedure and immediate morphological success with ≤ 50% residual stenosis (visual assessment) | Intraoperative
Device success, defined as exact deployment of the device according to the IFU (operator assessment) | Intraoperative
Procedural success, defined as the combination of technical success and device success | Intraoperative
Ankle-Brachial Index (ABI) at 6, 12 and 24 months (and prior to any reintervention) | 6, 12 and 24 months
Improvement of at least one Rutherford class at 6, 12 and 24 months (an prior to any reintervention) compared to the pre-procedure Rutherford classification. | 6, 12 and 24 months
Target Lesion Revascularization (TLR) and Target Vessel Revascularization (TVR) at 6, 12 and 24 months. | 6, 12 and 24 months
Limb salvage, defined as preservation of the treated limb with no need for any amputation at 6, 12 and 24 months. | 6, 12 and 24 months
Improvement of pain score at 6, 12 and 24 months compared to the pre-procedure score | 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (5):
  - Klinikum Hochsauerland, Karolinen-Hospital, Arnsberg
  - Knappschaftskrankenhaus Bottrop, Bottrop
  - SRH Klinikum Karlsbad-Langensteinbach GmbH, Karlsbad-Langensteinbach
  - Gefaesspraxis im Tal, München
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
- CHUV, Service de Chirurgie Vasculaire, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Lichtenberg M, von Bilderling P, Ranft J, Niemoller K, Grell H, Briner L, Saucy F, Rassaf T, Breuckmann F. Treatment of femoropopliteal atherosclerotic lesions using the ranger paclitaxel-coated balloon catheter: 12-month results from an all-comers registry. J Cardiovasc Surg (Torino). 2018 Feb;59(1):45-50. doi: 10.23736/S0021-9509.17.10261-2. Epub 2017 Oct 3. PMID 28980462